CLINICAL TRIAL: NCT00517205
Title: The Use of Non-contrast Helical Computerized Tomogram in Predicting Treatment Outcome of Upper Ureteric Stone by Extracorporeal Shock Wave Lithotripsy Using the Sonolith 4000+ Lithotripter
Brief Title: Study on 'The Use of Non-contrast Helical Computerized Tomogram in Predicting Treatment Outcomes of Upper Ureteric Stone by Extracorporeal Shock Wave Lithotripsy Using the Sonolith 4000+ Lithotripter'
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Other Study IDs: CRE-2004.309; HARECCTR0500008
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Ureteral Calculi
Keywords: upper ureteric stone
MeSH Terms: conditions — Ureteral Calculi; Ureterolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Non-contrast helical computerized tomogram (NCHCT)

SUMMARY:
The purpose of this research is to assess the role of non-contrast helical computerized tomogram in predicting the treatment outcome of upper ureteric stone by extracorporeal shock wave lithotripsy (ESWL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years old)
* With solitary upper ureteric stone (defined as ureter above the sacroiliac joint as seen on plain radiography) diagnosed by NCHCT *(* can have stones at the other site but the indexed stone is a solitary stone)
* Size 5 to 15 mm in the maximal diameter as measured from plain radiography.
* Planned for primary in-situ ESWL

Exclusion Criteria:

* Patient contraindicated for ESWL - active urosepsis, coagulopathy, pregnant lady etc
* Presence of percutaneous nephrostomy or ureteric stent
* Suspected distal obstruction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient suffered upper ureteric stone
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-10; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, Dr, Principal Investigator — Department of Surgery, Division of Urology, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China